CLINICAL TRIAL: NCT06271668
Title: Clinical Decision Support to Improve System Naloxone Co-prescribing
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 23-2356; R61DA057610 (NIH)
Record Dates: First submitted 2024-02-14; First posted 2024-02-22 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Medication Abuse; Harm Reduction; Opioid Overdose; Opioid Prescribing
MeSH Terms: conditions — Substance-Related Disorders; Harm Reduction; Opiate Overdose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical Decision Support (CDS): Naloxone Alert: Encounters where the naloxone clinical decision support (CDS) alert fired. CDS logic is programmed to fire alert when a provider places and order for a high-risk opioid analgesic prescription to a patient without an active naloxone prescription.
  High-risk prescription logic to trigger the Naloxone CDS:
  [(NOT 1 AND (2 AND AT LEAST 1 OF (3, 4, 5, 6))) AND 7 AND NOT 8]
  1. ACTIVE OR PENDED NALOXONE PRESCRIPTION ORDER
  2. OPIOID SCRIPT BEING PLACED CRITERIA
  3. DAILY Milligram Morphine Equivalent (MME) >=90 UNSIGNED ORDER
  4. DAILY MME >=90 EXISTING
  5. DIAGNOSIS OF OPIOID USE DISORDER
  6. DIAGNOSIS HISTORY OF OPIOID OVERDOSE
  7. PROVIDER LOGGED INTO ELLIGIBLE DEPARTMENTS
  8. DISCHARGE TO HOSPICE
  Interventions: Other: Naloxone Co-prescribing Clinical Decision Support (CDS)
- Usual Care: Control group of contemporary encounters where clinical decision support (CDS) is not active. Usual care.

INTERVENTIONS:
Other: Naloxone Co-prescribing Clinical Decision Support (CDS) — Clinical decision support in the form of an EHR-integrated, provider facing alert suggesting (a) the opioid medication order is considered high risk for overdose and (b) to nudge providers to add a naloxone prescription to the opioid prescription to mitigate risk in the event of an overdose.
  Groups: Clinical Decision Support (CDS): Naloxone Alert

SUMMARY:
The objective of this study is to evaluate the impact of a clinical decision support (CDS) alert to facilitate the co-prescribing of naloxone, an opioid overdose reversal agent, with high-risk opioid prescriptions. Prescribing naloxone with opioids is a best practice described in the 2022 US Center for Disease Control and Prevention (CDC) guidelines on opioid prescribing. The CDS can improve quality of care delivered by improving compliance with the guideline defined best practices. The project will compare CDS alert facilitated co-prescribing of naloxone with high-risk opioid prescriptions vs usual care to evaluate the effectiveness of the CDS alert for improving naloxone prescribing. The patients are not assigned to an intervention and will be receiving any changes in care as part of their routine medical care, rather than a specific intervention that is distinct from their usual medical care. The researchers hypothesize that the CDS alert will be acceptable to providers while increasing naloxone co-prescribing which will reduce the number of opioid overdoses in subsequent 6 months.

DETAILED DESCRIPTION:
Clinical decision support tools help clinicians make treatment decisions based on routinely collected data and offer a promising strategy to implement evidence-based practices for safe and effective pain management. This project will use clinical decision support tools embedded into electronic health records to help healthcare providers make treatment decisions that align with opioid prescribing guidelines from the Centers for Disease Control and Prevention (CDC). The project will also use information from prescription drug monitoring programs, insurance claims, and mortality data to evaluate patient outcomes. This research will evaluate how prescribing practices that align with CDC guidelines affect patient outcomes and whether clinical decision support tools provide an advantage over standard care practices for pain management.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving an opioid prescription at discharge from inpatient/ED or close visit in outpatient settings where the clinical decision support (CDS) is implemented

Exclusion Criteria:

* Patients <12 and >89 year of age
* Cancer diagnosis
* Hospice care/palliative care
* Sickle cell disease diagnosis
* Patients who arrived in error
* Patients who were triaged to obstetrics

Ages: 12 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Residents and visitors to the state of Colorado who seek healthcare within the University of Colorado Health (UCHealth) system.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of a high-risk opioid analgesic prescriptions receiving a co-prescription of naloxone | 18 months
  The number of high-risk opioid encounters where a naloxone prescription was written with the opioid divided by the total number of encounters where a high-risk opioid prescription was written.

SECONDARY OUTCOMES:
Clinical decision support (CDS) acceptance rate | 18 months
  The number of times providers accepted the Clinical decision support (CDS) suggestion and co-prescribed naloxone with a high-risk opioid divided by the total number of times a high-risk opioid prescription triggered the CDS alert.
Subsequent opioid overdose/poisonings rates | Six months after an encounter where the naloxone clinical decision support fired for the provider
  The number of patients who had a diagnosis of opioid overdose or poisoning in the six months following the index visit with a high-risk opioid prescribed.
Naloxone dispensed rate | In the 3 days after the naloxone prescription is written
  The number of patients who were dispensed a naloxone prescription divided by the number of naloxone prescriptions written.

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Hoppe, DO, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified quantitative EHR data utilized in this project will be housed on the National Addiction and HIV Data Archive Program (NAHDAP) website.
Supporting Information: Study Protocol
Time Frame: Data will be provided to NAHDAP after study results are published in peer-reviewed journals.
Access Criteria: Prior to downloading study data, the individual will have to register with the site and agree to a standard data use agreement.
URL: https://www.icpsr.umich.edu/web/pages/NAHDAP/index.html